CLINICAL TRIAL: NCT02125188
Title: Effects of Desmopressin on Blood Loss and the Quality of the Surgical Field During Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Department of anesthesiology, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: desmopressinFESS
Record Dates: First submitted 2014-04-21; First posted 2014-04-29 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Patients Undergoing Endoscopic Sinus Surgery
MeSH Terms: interventions — Deamino Arginine Vasopressin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Desmopressin (Experimental): Desmopressin 3ug/kg in saline 100ml ivdrip before surgery
  Interventions: Drug: Desmopressin
- saline (Placebo Comparator): saline 100ml ivdrip before surgery
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Desmopressin — Desmopressin 3ug/kg ivdrip before surgery
  Arms: Desmopressin
Drug: saline — saline 100ml ivdrip before surgery
  Arms: saline

SUMMARY:
Bleeding during functional endoscopic sinus surgery (FESS) is a challenge for both surgeons and anesthesiologists despite several measures available for improving the surgical field. This study was conducted to evaluate the effect of desmopressin on blood loss and the quality of the surgical field in FESS.

DETAILED DESCRIPTION:
Desmopressin, a synthetic analogue of vasopressin, has been employed as a non-transfusional treatment for hemophilia and von Willebrand's disease. Hemostatic effects of desmopressin include: 1) an increase in plasma factors through endogenous release of coagulation factor VIII, von Willebrand factor and tissue plasminogen activator; 2) an increase in platelet adhesiveness; and 3) a reduction in bleeding time. Randomized, double-blind studies have been performed on patients undergoing various types of surgical procedures. A study in patients undergoing orthognathic surgery showed a significant reduction in intraoperative blood loss and a study in patients undergoing lumbar fusion concluded that desmopressin was effective in reducing intraoperative blood loss. The purpose of this study was to investigate the effect of administration of desmopressin on intraoperative blood loss in patients undergoing FESS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II
* aged 18-60 years

Exclusion Criteria:

* Patients receiving anticoagulants
* medically important liver or kidney dysfunction
* significant heart disease
* allergy to Desmopressin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Blood loss | During Functional Endoscopic Sinus Surgery of each patient

SECONDARY OUTCOMES:
Quality of the surgical field using a scoring scale | During Functional Endoscopic Sinus Surgery of each patient
  The overall quality of the surgical field was assessed on a scoring scale adapted from Boezaart et al. The following are the scoring scale:
  0-1: No bleeding; excellent to outstanding surgical conditions; 2-3: Slight bleeding; surgery fairly easy. No stops for hemostasis and/or suctioning are required; 4-5: Slight bleeding; surgery mildly difficult. One stop for hemostasis and/or suctioning is required; 6-7: Moderate bleeding; surgery moderately difficult. Occasional stops for hemostasis and/or suctioning are required; 8-9: Moderate to severe bleeding; surgery very difficult. Multiple stops for hemostasis and/or suctioning are required; 10: Surgery terminated due to severe bleeding in the surgical field.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China